CLINICAL TRIAL: NCT07011264
Title: Development and Testing of BAJJAJJA: An Intervention to Promote Economic Empowerment and Health of Grandmothers Who Provide Primary Care for Grandchildren in Uganda
Brief Title: Economic Empowerment and Health Promotion of Uganda Grandmother-caregivers.
Acronym: BAJJAJJA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Makerere University (Other)
Responsible Party: Principal Investigator, Schola Matovu, PhD, RN, Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UUtah; 1K01TW012427-01A1 (NIH)
Record Dates: First submitted 2025-02-20; First posted 2025-06-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-05

CONDITIONS: Financial Burden; Health Behavior; Social Support
Keywords: NIH Stage Model; intervention testing; intervention development; physical challenges; mental challenges; financial stress; Ugandan grandmother-caregivers
MeSH Terms: conditions — Financial Stress; Health Behavior

STUDY DESIGN:
Intervention Model Description: The study will use the NIH Stage Model of behavioral intervention development following these stages:
  Stage IA: Intervention development (our preliminary work), Stage IB: Intervention refinement, modification, and adaptation and pilot testing (proposed/current study), Stage II: efficacy testing (future/subsequent study),
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Economic Empowerment and Health Promotion (Experimental): In this study, all 24 participants will engage in two intervention components constituting of an income generating activity (e.g. poultry farming) and health coaching (facilitated by visiting nurses).
  Interventions: Behavioral: The BAJJAJJA intervention

INTERVENTIONS:
Behavioral: The BAJJAJJA intervention — The BAJJAJJA intervention is composed of:
  The IGA COMPONENT which is intended to promote economic empowerment by improving household income based on available resources. The component will consist of a series of 1-hour sessions with 3 separate GMC participant groups (8 GMCs per group). Two IGA experts will lead these sessions, weekly for the first two months and later monthly for the remaining 10 months of the 12-month intervention period.
  The HEALTH COACHING COMPONENT will be informed by theChronic Disease Self-Management Education (CDSME) framework.54 This community-based, person-centered care model will be used to empower GMCs to manage their health through goal-setting, problem-solving, and chronic disease self-monitoring. I (PI) will leverage the community networks that I developed during my preliminary work to (1) recruit interventionists (two nurses) and (2) ensure their adequate training and adherence to the intervention manuals and procedures.

SUMMARY:
Background:

There are an estimated 163 million children worldwide who are under the care of their grandparents or other relatives. In Uganda, social determinants of health (i.e., poverty, wars, and maternal and perinatal conditions) threaten the middle generation (age 15-49) and leave older adults, especially grandmothers (Bajjajja), to become the safety net. Yet, in this region, knowledge about effective interventions that support the health and wellbeing of these GMCs is limited to nonexistent. As such, Dr. Matovu proposes to refine, adapt, and test her BAJJAJJA intervention that she developed.

Specific Aims:

Dr. Matovu will achieve this goal through three Specific Aims:

1. Refine and adapt the BAJJAJJA intervention components through a collaborative and iterative feedback process with a diverse community group of 18 members;
2. Test the feasibility, acceptability and preliminary efficacy of the BAJJAJJA intervention in improving economic and health outcomes among 24 Ugandan GMCs; and
3. Explore the barriers and facilitators to (3a) maintenance of the BAJJAJJA individual intervention benefits and (3b) sustainability of the income generating activity at 6 months post-intervention.

This innovative study will utilize a community-engaged approach that emphasizes the meaningful involvement of community partners to develop an intervention that targets GMCs. Her outcomes will support her future efficacy clinical trial to test a novel multi-component and community-engaged BAJJAJJA intervention to promote the mental, physical, and economic wellbeing of GMCs.

DETAILED DESCRIPTION:
SIGNIFICANCE Caring for children is complex in the best of circumstances. Grandparents take on primary caregiving responsibility when parents are unavailable or unable to rear their children. In sub-Saharan Africa, prevailing reasons for grandparent-caregiving include parental illness/death due to AIDS and other infectious diseases and socioeconomic factors such as chronic poverty.1-8 Although sub-Saharan Africa has seen reductions in new HIV infections compared to other regions, it remains the most affected worldwide. Of the estimated 13.4 million orphans created by the HIV/AIDS epidemic, more than 80% live in sub-Saharan Africa,9 and grandmothers often step forward to care for orphaned children.1-8,10 Older grandmothers (bajjajja), some of whom are living with HIV, bear the additional responsibility of caring for children who may be infected with HIV and/or have other special needs. Dr. Matovu's research will focus on Uganda, a country with a long history of HIV cases,11 and older grandmother-caregivers (GMCs) who often become the primary caregivers for their grandchildren. Without the safety net provided by GMCs, Uganda could face a public health crisis.

Grandparent-Caregiving Phenomenon:

The plight of GMCs has been documented by exploratory studies in Uganda as it relates to social determinants of health (SDoH) such as wars and the early years of the HIV epidemic.1-9 Many of these studies highlighted the challenges and few rewards of caregiving as experienced by Ugandan GMCs. However, these studies did not explore GMCs' perception of their role, the intricate familial restructuring or decision-making involved in caring for grandchildren affected by HIV/AIDS, or the impact of caregiving on mental and physical health of these older adults. These gaps motivated me to explore the grandparent-caregiving phenomenon as experienced by older Ugandan grandparents. From a qualitative study of 32 Ugandan GMCs, the PI developed the GRAndparent-CarEgiving (GRACE) model, a substantive theory12,13 that offers a theoretical explanation of the caregiving experience and role as reported by GMCs (publication in review). The findings from this foundational research begun to fill the prior gaps in knowledge and further established an understanding of key concepts, such as symptom experience,14 loss,15 perceived rewards, stress, and coping16,17 as experienced by GMCs. Alongside corroborating positive aspects of caregiving from prior studies,8,9 the foundational research revealed overwhelming caregiver stress. Grandparents reported physical, emotional, social, and, most prevalently, financial burdens that impacted their abilities to adequately provide for themselves, their grandchildren, and other family members, such as aging spouses and parents.

The proposed intervention will target GMCs' primary support needs: financial and health-related wellbeing. A handful of descriptive caregiver studies in sub-Saharan Africa explored the impact of caregiving on younger family caregivers (~39 to 48 years of age) and reported extensive caregiver burden, poor nutritional status, and potential adverse health outcomes, such as cardiovascular disease and depression.18,19 The paucity of research in sub-Saharan Africa, particularly in Uganda, contrasts with the extensive research in North America, showing the negative impact of caregiving on the physical and mental health of GMCs.20-40 Additionally, there are a few intervention studies in Central and East African that focus on women's empowerment41,42 and AIDS orphans and their families.43-46 While highlighting the challenges experienced by the younger caregiver cohort and orphans, findings from these studies may not directly translate to the specific needs of an aging population of GMCs in Uganda. Grandmothers are particularly vulnerable to age-related poor health outcomes and chronic socioeconomic stressors that may be further exacerbated by caregiving.24, 29,32 These women are often responsible for the wellbeing of their families, especially when diseases and other SDoH negatively impact the productive and reproductive age group (15-49).17 Therefore, compromised health among GMCs can potentially affect a whole family, leading to increased adverse social, health, and economic community outcomes. The next logical step in advancing this research among GMCs is to refine and adapt an innovative and multi-component intervention, BAJJAJJA: Building A Joint Action for JaJJAs, and test its feasibility, acceptability, and preliminary efficacy. The PI proposed research will be the first known study to test a multi- component intervention geared toward the unique needs of GMCs in Uganda.

Scientific Premise and Theoretical Underpinnings: the intervention is informed by Pearlin's47 interpretation of the stress process and Lazarus and Folkman's transactional model of stress and coping.48 The PI's preliminary research enabled me to contextualize the application of these two theories to the specific stressors experienced by older GMCs in Uganda.14-17,49 It is essential that the investigators address these stressors through culturally appropriate interventions. The proposed intervention will, therefore, focus on two of the most salient stressors: financial and health challenges. The BAJJAJJA intervention is comprised of two components: (1) an income generating activity (IGA) and (2) nurse-led health coaching. These intervention components align with two of the social support typologies proposed by House:50 instrumental/tangible (earnings from the IGA) and informational (health coaching). Providing social support in these categories has potential to reduce the effects of stress and improve the financial and health outcomes of GMCs.

INNOVATION The BAJJAJJA intervention is the first (that the investigators know of) to explore the effectiveness of an IGA and health coaching in promoting household income and health among Ugandan GMCs. The proposed study is also the first (that the investigators know of) in Uganda to utilize a community-engaged approach to emphasize the meaningful involvement of community partners to inform intervention development for GMCs. Engaging community partners in all study phases is critical to allow for a community-informed development, validation, and evaluation of a culturally relevant, sustainable intervention. The BAJJAJJA intervention aligns with the Uganda National Council for Science and Technology's priorities to develop regulations that will soon require all studies conducted with human subjects to involve a level of community engagement.51 Results of the proposed study have the potential to (1) advance gerontological and grandparent-caregiving research by testing interventions that address SDoH affecting an aging population, (2) improve economic and health behavior outcomes, and (3) advance the PI's program of research by informing a subsequent R01 efficacy trial.

APPROACH Study Objective: Following the NIH Stage Model,66 the proposed study aims to (1) use a community-engaged approach to engage a diverse group of community members in the refinement and adaptation of the BAJJAJJA intervention (AIM 1); (2) test the intervention's feasibility, acceptability, and preliminary efficacy (AIM 2); and (3) explore the barriers and facilitators to the long-term maintenance of the intervention (e.g., physical activity level and frequency) and sustainability of the IGA activities (e.g., accessing of external supports such as community resources) at 6 months post-intervention (AIM 3).

THE BAJJAJJA INTERVENTION:

There is growing evidence that multi-component economic empowerment and health promoting interventions, like the BAJJAJJA intervention, can be feasibly scaled to national and regional levels.41-45 The IGA COMPONENT is intended to promote economic empowerment by improving household income based on available resources. Informed by CAB members,49 I adapted the USAID IGA guidelines53 to develop an IGA manual. Working closely with Dr. Namisango, an economist and K01 Advisor, a budget will be established to provide direct funds for the IGA project. The intervention will consist of a series of 1-hour sessions with 3 separate GMC participant groups (8 GMCs per group). Two IGA experts will lead these sessions, weekly for the first two months and later monthly for the remaining 10 months of the 12-month intervention period. In the first phase, the experts will assist the group in determining governance, communication, roles, responsibilities, and how they plan to steward their funds. The second phase will involve education on IGA topics, such as market assessment, cost-benefit analysis, production and marketing, bookkeeping, and market niche/materials, to enhance knowledge about management, entrepreneurship, sustainability planning, and awareness of community resources to support the IGA post- intervention.49 As informed by the preliminary work, the 3 GMC groups may identify others (e.g., older grandchildren or community members) to assist in IGA tasks, such as feeding livestock. A formal caretaker may also be hired to assist the GMCs with heavier tasks due to physical and mobility challenges. Identified helpers will be invited to join select sessions to increase their knowledge of animal husbandry. The final phase will be guided by elements of implementation fidelity.68,81

The HEALTH COACHING COMPONENT will be informed by the Chronic Disease Self-Management Education (CDSME) framework.54 This community-based, person-centered care model will be used to empower GMCs to manage their health through goal-setting, problem-solving, and chronic disease self-monitoring. I (PI) will leverage the community networks that I developed during the preliminary work to (1) recruit interventionists(two nurses) via established networks and or newspaper advertisements and (2) ensure their adequate training and adherence to the intervention manuals and procedures. I will lead a 2-day training workshop with the two interventionists on the content, delivery, and format of the CDSME health-topic modules (e.g., pain management, nutrition, physical activity, medication use, sanitation, and emotions) and motivational interviewing (MI) techniques. Interventionists will then (1) conduct participant assessments and monitor health indicators at three time points (baseline, 12 months, and post-intervention [18 months]), and (2) facilitate the group health coaching sessions (each 1.5 hours long), weekly for the first two months and later monthly for the next ten months using the developed coaching materials and MI. Published randomized controlled trials suggest that using MI with older adults can lead to modifications to health-related behaviors and works well in group settings; further, MI promotes empowerment and engagement in managing and improving health outcomes.55-59 Interventionists will employ the four-phase group MI model: (1) engaging the group (e.g., developing working relationships, norms within the group, and guidelines); (2) exploring participants' perspectives (e.g., on their values, health and health goals, barriers and issues, and ambivalence); (3) broadening perspectives (e.g., generating potential options for change, identifying strategies to overcome barriers); and (4) moving into action (e.g., setting goals, planning and implementing changes that participants believe will improve their lives).59

Specific Aim 1: To refine and adapt the BAJJAJJA intervention components through a collaborative and iterative feedback process with a diverse community group of 18 members.

Sample and Setting: AIM 1 will focus on refining the BAJJAJJA intervention, including study measures and training materials.49 In this aim, 18 participants will be recruited from rural areas around Masaka, Luwero, or Lugazi, regions historically most affected by HIV/AIDS and sociopolitical factors. Participants will include elected local council (LC) leaders (n = 3), healthcare professionals (n = 3; 2 nurses from local health centers and 1 village health team member),60 IGA experts (n = 2), and GMCs (two focus groups of five participants each, n = 10 total). Participants will be recruited if they live or work in adjacent villages of the research site and can speak English and or Luganda (commonly spoken languages). The GMCs will be > 50 years, younger GMCs will be excluded (see Eligibility Criteria). Participants will be identified by LC leaders or referred by other participants using a snowball sampling technique.61 Methods: Data Collection: The investigators will conduct two phases of data collection: 1) Verification and 2) Cognitive Interviewing. First, the investigators will divide participants into subgroups (1: LCs, 2: health team, and 3: IGA experts) and two GMC Focus Groups. During the Verification Phase, the investigators will engage Subgroups 1, 2, and 3 in separate discussions related to their role in the community and the intervention. Subgroup 1 will provide feedback on the welfare and community activity/organization aspects of the intervention, such as how to secure a site for the IGA or management of any conflict that may arise in the GMC groups during AIM 2. Subgroup 2 will provide feedback on the health coaching components, and Subgroup 3 will offer feedback on the IGA components.

Data will be collected via semi-structured interviews in this phase. In the Cognitive Interviewing Phase, the investigators will conduct discussions with the two GMC focus groups using a group-based cognitive interviewing62 technique for another round of refinement. The two focus group sessions will last 1.5 hours each. This phase will also ensure a robust and unbiased approach to data source triangulation, allowing for community-informed validation, evaluation, and development of a culturally relevant intervention. Semi-structured interview guides with prompt questions will ensure an exhaustive exploration of the participants' perspectives on the intervention components verified by the subgroups in the previous phase. Field notes will be made, and focus group discussions audio-recorded, transcribed, and transferred into Atlas.ti software for analysis. If needed, the investigators may increase the number of GMC focus groups to promote member checking63 or achieve theoretical saturation.64 Data Analysis: The semi-structured interview data from both the Verification and Cognitive Interviewing Phases will be analyzed using thematic analysis and evaluation of verbalized cognitive processes. In the Verification Phase, qualitative data analysis will follow the six steps of thematic analysis:65 (1) familiarization (thorough review of all transcribed data); (2) coding (deconstructing data to clusters/units/codes of meaning); (3) generating themes (reviewing created codes to identify patterns); (4) reviewing themes (ensuring that themes are useful and accurate representations of the data); (5) defining and naming themes; and (6) writing up the analysis. Key themes will be identified to examine the quality and content of the intervention components and identify elements that may need to be refined to improve future intervention iterations. In the Cognitive Interviewing Phase, the investigators will analyze the GMCs' cognitive processes by (1) producing summaries (describing how GMCs understood the question as well as how they came up with their responses, taking into account any relevant events or experiences and any challenges they encountered); (2) comparing data across the two focus groups by identifying and mapping common themes and different perspectives; and (3) reaching conclusions (determining and explaining the performance of a question as it functions within the group context). This data analysis process will be iterative and reductive. To ensure analytic rigor for AIM 1, two coders (PI and Research Assistant) will independently code the data, and a third party (a mentor) will arbitrate consensus. At the conclusion of this aim, the investigators will have refined the BAJJAJJA intervention components and adapted them following the NIH Stage Model and ready for Stage 1B: Feasibility and Pilot Testing.

Specific Aim 2: To test the feasibility, acceptability, and preliminary efficacy of the BAJJAJJA intervention in improving economic and health outcomes among 24 Ugandan GMCs.

Sample and Setting: The investigators will recruit 24 Ugandan GMCs who are (a) > 50 years (considering the average reproductive age range in Uganda of 15-49 years),67 (b) Luganda-speaking (commonly spoken language), (c) primary caregivers for at least one minor grandchild (< 18 years) for > 6 months, and (d) able to perform activities of daily living (e.g., cooking, bathing) without assistance. The investigators will exclude grandmothers who cohabitate with their adult children. Grandmothers will be initially referred by the CAB or participants in AIM 1 and later by snowball sampling.61 Three groups of 8 GMCs will be formed from adjacent villages. The PI's preliminary study49 substantiated that GMCs are willing to convene at locations convenient to all (e.g., neighboring schools) and would usually walk to the research site.

Methods: AIM 2 will utilize a mixed methodology with a quasi-experimental design. The investigators will collect qualitative and quantitative data to assess the feasibility, acceptability, and preliminary efficacy of the intervention.

Intervention Delivery: Participants will be assigned to one of the three GMC groups to optimize group dynamics. The BAJJAJJA intervention will be delivered in two phases over a 12-month period: weekly for the first 2 months and then monthly for the following 10 months. Sessions will last 3 hours (30 min of pre- and post-session activities, 1.5 hours of the health component, and 1 hour of the IGA component).

Implementation Fidelity: Intervention delivery will be guided by the elements of implementation fidelity:

adherence to intervention design, dosage and exposure, quality of delivery, and participant responsiveness.68,81 Since I will not be involved in intervention delivery, I will rate fidelity to reduce bias. I will 1) attend all intervention sessions, 2) supervise and give feedback to the interventionists on module delivery and content, and 3) perform weekly and later monthly IGA site visits and behavioral observations to ensure adherence to the prescribed activities and practices from the educational modules and intervention manual. I will also ensure interventionists' competence in content delivery. Other fidelity measurement methods and tools include audio recordings of sessions, the MI Fidelity checklist,69 a modified quantitative fidelity instrument and checklist,70,81 and self-report fidelity measures that ask interventionists to indicate whether they implemented specific components of the intervention protocol.

Feasibility and Acceptability: Feasibility and acceptability data will be captured using frequencies and percentages. Feasibility will be assessed based on the number and percentage of participants who attend the intervention sessions. Attendance rosters will track who attends and for how long. Informed by standard guidelines,71 the intervention will be considered feasible if at least 70% of the invited participants attend at least 8 of 12 scheduled group sessions. The investigators will estimate recruitment and retention rates and document reasons for attrition. Descriptive statistics will be reported for measures completed over the three time points (baseline, 12 months, and post-intervention). Acceptability will be summarized based on an average score from a satisfaction survey and qualitative interviews. Using a 5-point Likert scale, participants will be asked to rate their satisfaction with the intervention format and facilitators (affective attitude), the amount of effort required to participate (burden of recommended exercises), and the extent to which they understand the intervention and how it is intended to work (intervention coherence). A professional transcriber will prepare focus group data from the audio recordings of the intervention sessions.

Data Collection: The investigators will collect demographic data using forms tailored to the Ugandan setting. Health indicators have been selected to map onto the conceptual model. Interviewer-administered survey data will be collected using survey instruments. Clinical data, including body mass index, blood pressure, and blood glucose, and Interviewer-administered survey data will be collected at baseline, 12 months, and 6 months post-intervention (18 months) by nurses. Upon completion of AIM 2, the investigators will conduct focus group discussions using semi-structured interviews with the three GMC groups to gather feedback on (1) perceived health knowledge, behavior change, motivations, skills, and attitudes towards health management and (2) ongoing barriers to implementation and suggestions for component modification.

Data Analysis: Quantitative: Working closely with Dr. Sheng, I will summarize quantitative metrics using descriptive statistics. The investigators will graph and visually inspect changes from baseline to follow-up on feasibility, acceptability, intervention impact measures, and preliminary efficacy measures on economic and health outcomes. The investigators will also examine differences in mean pre- and post-intervention scores that will inform future power analyses. No inferential statistics are planned due to the small sample size and the preliminary nature of the proposed project. Qualitative: Transcribed qualitative data will be analyzed using thematic analysis as described in AIM 1. In addition, the investigators will develop a codebook, which will include a list of codes with their definitions, to structure interpretation of text. In the first cycle of analysis, the investigators will utilize a deductive approach to review the priori structural codes from the conceptual model and existing knowledge. The integration process of both quantitative and qualitative data will involve creating a crossover visualization79 to map out the results. When this aim is completed, the investigators will have established whether the intervention is feasible, acceptable, and effective for improving economic and health outcomes.

Specific Aim 3: To explore the barriers and facilitators to (3a) maintenance of the BAJJAJJA individual intervention benefits (e.g., physical activity level and frequency) and (3b) sustainability of the IGA activities (e.g., grandmothers' accessing external supports such as community resources) at 6 months post-intervention.

Sample and Setting: At 6 months post-intervention, the 24 GMCs from AIM 2 will be interviewed to provide their insights on the long-term maintenance or continuation of behavior related to targeted individual outcomes (e.g., consistent physical activity) (3a) and (2) sustainability of the IGA process and activities (e.g., accessing of external supports such as community IGA resources) (3b). Methods: Data Collection: The investigators will use a mixed methods approach to collect data on health measures and clinical outcomes similar to those used in AIM 2. Qualitative Data: I (PI) will conduct one-on-one semi structured, in-depth interviews with the 24 GMCs from AIM 2 to explore challenges related to health behavior change, motivations, and changes in perceived knowledge, skills and attitudes, and facilitators of and barriers to sustaining IGA activities. Quantitative Data: Survey measures and clinical data (e.g., body mass index, blood pressure, and blood glucose) collected as part of AIM 2 (baseline and 12 months), will be examined with a lens for sustainability and maintenance.

Data Analysis: Qualitative data analysis will follow procedure outlined in AIM 1 and 2. Quantitative data analysis will again use descriptive statistics as outlined in AIM 2. While no pre-specified hypotheses are planned, the investigators will describe associations between individual demographic, social-economic, and other factors to interventional benefits and sustainability to understand potential barriers and facilitators for a larger-scale research project. For mixed methods, a data integration process will involve creating a crossover visualization79 to map out the results.

POTENTIAL PITFALLS AND ALTERNATIVE APPROACHES [AIMS 1-3] I have identified potential barriers to the successful completion of AIMS 1-3 as they relate to 1) recruitment, 2) retention, 3) CAB member and participant fatigue, and 4) intervention component challenges. I have established a strong, interdisciplinary mentoring team and community networks and partnerships through the preliminary work that will facilitate effective resolutions to overcome barriers as follows: 1) To address potential recruitment delays, I will partner with CAB members to expand recruitment to adjacent villages and, as needed, access a previously established participant registry (see Recruitment and Retention Plan). 2) To optimize retention, the PI will adhere to the Retention Plan, which includes participant incentives, maintaining regular participant engagement (i.e., follow-up calls, home visits). Also, I will provide the option of holding interviews/meetings near participants' residences and offer flexible meeting times. 3) To reduce potential fatigue, the investigators will regularly reevaluate the frequency and duration of meetings/sessions, ensuring flexibility and avoiding attrition. 4) To identify participant concerns or potential barriers to achieving planned IGA or health intervention goals, such as concerns related to health modules, an assessment will be incorporated into the monthly intervention sessions. Throughout the duration of the proposed study, I will regularly consult with the mentorship team to troubleshoot potential pitfalls and devise alternative approaches to resolve them.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

* Female, aged 50 years or older (reflecting the post-reproductive age range in Uganda)
* Luganda-speaking (commonly spoken language).
* Primary caregiver of at least one minor grandchild (under 18 years) for more than six months
* Able to independently perform activities of daily living (e.g., cooking, bathing)

Exclusion Criteria:

Participants will be excluded if they:

* Are cohabitating with their adult children
* Are grandmothers under the age of 50

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Mental and Physical Health: Short Form Health Survey - 12-Item Version (SF-12) | Baseline, 12-months, and 6- months post-intervention (18- months)
  12 item self-reported outcome measure that assesses the impact of health on an individuals everyday life. It addresses 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role and mental health.
  Scoring Range: Physical Component Summary (PCS) & Mental Component Summary (MCS): typically ranges from 0 to 100 Interpretation: Higher scores on both the PCS and MCS indicate better health outcomes (better physical functioning and mental well-being).
Caregiver Strain: Zarit Burden Interview (ZBI) | Baseline, 12-months, and 6- months post-intervention (18- months)
  13 questions to measure caregiver strain in at least one of the following domains: Financial, Physical, Psychological, Social, and Personal.
  Scoring Range: The standard 22-item version of the Zarit Burden Interview has a total score range from 0 to 88. Each item is scored on a scale from 0 (Never) to 4 (Nearly Always).
  Interpretation: Higher scores indicate a worse outcome, meaning greater caregiver strain or burden. Lower scores suggest less perceived burden.
Self-Eﬃcacy: Short Form of General Self-Eﬃcacy Scale (GSE-6) | Baseline, 12-months, and 6- months post-intervention (18- months)
  6-item Short Form of General Self-Eﬃcacy Scale assesses a sense of perceived self-eﬃcacy aimed to predict coping and adaptation with stress
  Scoring Range: The 6-item short form has a total score range from 6 to 30. Each item is typically rated on a 5-point Likert scale from 1 (Not at all true) to 5 (Exactly true).
  Interpretation: Higher scores indicate a better outcome, meaning greater self-efficacy. Lower scores suggest less confidence in one's ability to cope with challenges or exert control over life circumstances.
Economic Empowerment: Women's Empowerment in Agriculture Index (WEAI) | Baseline, 12-months, and 6- months post-intervention (18- months)
  12 indicators including, autonomy in income, self-eﬃcacy, ownership of land and other assets, access to and decisions on credit, control over use of income, work balance, group membership, etc.
  Scoring Range: The Women's Empowerment in Agriculture Index score ranges from 0 to 1.
  Interpretation: Higher scores indicate a better outcome, meaning greater empowerment in agriculture-related domains. A score of 1.0 represents full empowerment, while a score closer to 0 indicates low empowerment.
Social Support: Duke-University of North Carolina Functional Social Support Questionnaire (Duke-UNC FSSQ) | Baseline, 12-months, and 6- months post-intervention (18- months)
  The Duke-University of North Carolina Functional Social Support Questionnaire measures a person's satisfaction with the functional aspects of social support. Scoring Range: The Duke-University of North Carolina Functional Social Support Questionnaire is scored on a 5-point Likert scale ranging from 1 (Much less than I would like) to 5 (As much as I would like). The total score ranges from 8 to 40.
  Interpretation: Higher scores indicate a better outcome, meaning greater perceived functional social support. Lower scores suggest less perceived support.
Food Insecurity & Household Income: Household Food Insecurity Access Scale (HFIAS) | Baseline, 12-months, and 6- months post-intervention (18- months)
  9-item instrument that addresses 3 domains of core experiences: uncertainty or anxiety about food supply; insuﬃcient food quality; and insuﬃcient food intake and its physical consequences
  Scoring Range: The Household Food Insecurity Access Scale is scored from 0 to 3 based on frequency of occurrence:
  0 = Never
  1. = Rarely (once or twice in the past four weeks)
  2. = Sometimes (three to ten times)
  3. = Often (more than ten times) Total score range: 0 to 27
  Interpretation: Higher scores indicate a worse outcome, meaning greater household food insecurity. Lower scores reflect better food access and food security.
Readiness to Change: Readiness to Change Questionnaire (RCQ) | Baseline, 12-months, and 6- months post-intervention (18- months)
  2-item to assess where individuals are in the cycle of change to inform goal setting, actions, and determine the best strategies.
  Scoring Range: The Readiness to Change Questionnaire is divided into three response subscales: Precontemplation, Contemplation. Action. Each item is scored from 1 (Strongly disagree) to 5 Scoring Range: The Readiness to Change Questionnaire is divided into three response subscales: Precontemplation, Contemplation. Action. Each item is scored from 1 (Strongly disagree) to 5 (Strongly agree).
  Interpretation:
  There is no single total score for the Readiness to Change Questionnaire; rather, the highest subscale score indicates the participant's current stage of readiness to change. Higher scores in the "Action" subscale suggest a better outcome, reflecting greater readiness to change.
  Higher scores in the Precontemplation stage indicate lower readiness (worse outcome in terms of behavior change).Contemplation is a middle stage of ambivalence or consideration.

SECONDARY OUTCOMES:
Feasibility & Acceptability: Demographic and Clinical Data Form | Baseline, 12-months, and 6- months post-intervention (18- months)
  Assess items which may contribute to health disparity, stress, and participation in healthy lifestyle behaviors (income, marital status, grandchildren, education level attained, etc.).
Sustainability & Maintenance: Semi-structured & structured questionnaires | Baseline, 12-months, and 6- months post-intervention (18- months)
  To explore barriers and facilitators to maintenance and sustainability of targeted individual health and IGA outcomes.
Fidelity Monitoring | Baseline, 12-months, and 6- months post-intervention (18- months)
  # of participants: screened for eligibility; assessed at timepoints, participated in intervention sessions.

OTHER OUTCOMES:
Weight | Baseline, 12-months, and 6- months post-intervention (18- months)
  * Measurement Method: Participants' weight will be measured using a calibrated digital scale.
  * Units: Kilograms (kg)
  * Procedure: Participants will be asked to remove shoes and any heavy clothing. The weight will be recorded to the nearest 0.1 kg.
Height | Time Frame: Baseline, 12-months, and 6- months post-intervention (18- months)
  * Measurement Method: Height will be measured using a stadiometer.
  * Units: Meters (m)
  * Procedure: Participants will stand upright without shoes, with their back against the stadiometer, and height will be recorded to the nearest 0.1 cm (then converted to meters).
Body Mass Index (BMI) | Time Frame: Baseline, 12-months, and 6- months post-intervention (18- months)
  o Calculation Method: BMI will be calculated using the formula: BMI = Weight (kg) / [Height (m)]²
  * Units: kg/m²
  * Interpretation: BMI values will be categorized according to WHO guidelines (e.g., underweight, normal, overweight, obese).
Blood Pressure | Time Frame: Baseline, 12-months, and 6- months post-intervention (18- months)
  * Measurement Method: Blood pressure will be measured using an automated digital sphygmomanometer.
  * Units: Millimeters of mercury (mmHg)
  * Procedure: Measurements will be taken on the participant's upper arm after 5 minutes of rest, in a seated position. Two readings will be taken at 1-minute intervals, and the average of the two readings will be used for analysis.
  * Reported Values: Systolic and diastolic blood pressure (e.g., 120/80 mmHg)
Blood Glucose | Time Frame: Baseline, 12-months, and 6- months post-intervention (18- months)
  * Measurement Method: Capillary blood glucose will be measured using a point-of-care glucometer (finger prick test).
  * Units: Milligrams per deciliter (mg/dL) or millimoles per liter (mmol/L), depending on local standards.
  * Procedure: Participants will be tested under fasting or random conditions, which will be recorded. Measurements will follow device-specific protocols.
  * Reported Values: Single value per participant, interpreted based on ADA/WHO clinical guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah College of Nursing, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
DISSEMINATION PLAN
  The investigators are interested in sharing of data generated by this project with others such as the general population and community of scientists interested in family caregiving, gerontology, and women economic empowerment interventions.
  REPORTING THROUGH CLINICALTRIALS.GOV Results from the developed intervention will be submitted to ClinicalTrials.gov no later than 1 year of the trial's primary completion date. Publications will be submitted to the National Library of Medicine PubMed Central website after acceptance to ensure dissemination of findings to the public.
  CONSENT DOCUMENTATION To inform study participations as to how the data of the proposed trial will be disseminated, the informed consent document will include a specific statement that the clinical trial information will be posted at ClinicalTrials.gov.
  INSTITUTIONAL POLICIES The University of Utah and Makerere University Co
Supporting Information: Study Protocol
URL: https://reporter.nih.gov/search/xHobiVLiPU68u-6wSogmsA/project-details/11052906

REFERENCES:
- [Background] Matovu S, Dawson-Rose C, Weiss S, Wallhagen M. "Thoughts Can Kill You": Characterization of Mental Health Symptoms by Ugandan Grandparent-Caregivers in the HIV/AIDS Era. Issues Ment Health Nurs. 2019 May;40(5):391-398. doi: 10.1080/01612840.2018.1553001. Epub 2019 Mar 27. PMID 30917054
- Available data/document: Study Protocol — https://reporter.nih.gov/search/xHobiVLiPU68u-6wSogmsA/project-details/11052906